CLINICAL TRIAL: NCT00677378
Title: Capsaicin-sensitive Transient Receptor Potential Vanilloid One (TRPV1) and Tyrosine Kinase (TrkA) Receptor Expression in Children With Retrosternal Pain
Brief Title: Transient Receptor Potential Vanilloid One (TRPV1) Receptor Expression in Children With Retrosternal Pain
Acronym: TRPV1
Status: Completed | Type: Observational
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Manu Sood, Chief, Associate Professor, Medical College of Wisconsin
Other Study IDs: CHW 06/34
Record Dates: First submitted 2008-05-09; First posted 2008-05-14 (Estimated); Last update posted 2015-10-22 (Estimated); Status verified 2015-10

CONDITIONS: Epigastric Pain; Retrosternal Pain; Esophagitis; Gastrointestinal Symptoms
Keywords: TRPV1; Nerve growth factor; Capsaicin; TrkA; Retrosternal pain; Epigastric pain; Esophagitis; Gastrointestinal symptoms
MeSH Terms: conditions — Esophagitis; Hereditary Sensory and Autonomic Neuropathies

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — We are collecting a single mucosal biopsy during an endoscopy procedure.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- EXPERIMENTAL: Children undergoing an endoscopy for retrosternal chest pain, epigastric pain, regurgitation, heart burn or dyspepsia.
- CONTROL: Children undergoing an endoscopy for reasons not stated in the experimental group condition (i.e. celiac disease, rectal bleeding, polyps, weight loss, malabsorption).

SUMMARY:
We would like to evaluate the changes in nerve innervation and TRPV1 receptor expression along with microscopic changes associated with heart burn and abdominal pain

DETAILED DESCRIPTION:
Approximately 5% of children between 10-17 years of age report symptoms of heart burn, epigastric pain or regurgitation. This study will evaluate the changes in nerve innervation and TRPV1 receptor expression in children having upper endoscopy for evaluation of heart burn and abdominal pain.

ELIGIBILITY:
Inclusion Criteria:

* Retrosternal and/or epigastric pain and esophagitis
* Retrosternal and/or epigastric pain but no macroscopic or microscopic esophagitis
* Gastrointestinal symptoms such as diarrhea, regurgitation, rumination, vomiting, feeding aversion, non-organic failure to thrive, celiac disease with no macroscopic or microscopic esophageal inflammation

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children undergoing an endoscopy procedure for gastrointestinal symptoms and chest pain or reasons other than those listed in the exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 77 (Actual)
Dates: Start 2006-12; Primary Completion 2014-12 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
To characterize the TRPV1 expression in the esophageal mucosa of children with esophagitis and to correlate the TRPV1 expression with severity of mucosal inflammation and microscopic changes. | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Manu Sood, MD, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Medical College of Wisconsin, Milwaukee, Wisconsin, United States

REFERENCES:
- [Background] Nelson SP, Chen EH, Syniar GM, Christoffel KK. Prevalence of symptoms of gastroesophageal reflux during childhood: a pediatric practice-based survey. Pediatric Practice Research Group. Arch Pediatr Adolesc Med. 2000 Feb;154(2):150-4. doi: 10.1001/archpedi.154.2.150. PMID 10665601
- [Background] El-Serag HB, Bailey NR, Gilger M, Rabeneck L. Endoscopic manifestations of gastroesophageal reflux disease in patients between 18 months and 25 years without neurological deficits. Am J Gastroenterol. 2002 Jul;97(7):1635-9. doi: 10.1111/j.1572-0241.2002.05820.x. PMID 12135011
- [Background] Carlsson R, Galmiche JP, Dent J, Lundell L, Frison L. Prognostic factors influencing relapse of oesophagitis during maintenance therapy with antisecretory drugs: a meta-analysis of long-term omeprazole trials. Aliment Pharmacol Ther. 1997 Jun;11(3):473-82. doi: 10.1046/j.1365-2036.1997.00167.x. PMID 9218069
- [Background] Sarkar S, Hobson AR, Furlong PL, Woolf CJ, Thompson DG, Aziz Q. Central neural mechanisms mediating human visceral hypersensitivity. Am J Physiol Gastrointest Liver Physiol. 2001 Nov;281(5):G1196-202. doi: 10.1152/ajpgi.2001.281.5.G1196. PMID 11668028
- [Background] Mehta AJ, De Caestecker JS, Camm AJ, Northfield TC. Sensitization to painful distention and abnormal sensory perception in the esophagus. Gastroenterology. 1995 Feb;108(2):311-9. doi: 10.1016/0016-5085(95)90055-1. PMID 7835571
- [Background] Cervero F. Visceral hyperalgesia revisited. Lancet. 2000 Sep 30;356(9236):1127-8. doi: 10.1016/S0140-6736(00)02750-1. No abstract available. PMID 11030288
- [Background] Faussone-Pellegrini MS, Taddei A, Bizzoco E, Lazzeri M, Vannucchi MG, Bechi P. Distribution of the vanilloid (capsaicin) receptor type 1 in the human stomach. Histochem Cell Biol. 2005 Jul;124(1):61-8. doi: 10.1007/s00418-005-0025-9. Epub 2005 Jul 22. PMID 16041554
- [Background] Cervero F, Laird JM. Understanding the signaling and transmission of visceral nociceptive events. J Neurobiol. 2004 Oct;61(1):45-54. doi: 10.1002/neu.20084. PMID 15362152
- [Background] Yiangou Y, Facer P, Dyer NH, Chan CL, Knowles C, Williams NS, Anand P. Vanilloid receptor 1 immunoreactivity in inflamed human bowel. Lancet. 2001 Apr 28;357(9265):1338-9. doi: 10.1016/s0140-6736(00)04503-7. PMID 11343743
- [Background] Chan CL, Facer P, Davis JB, Smith GD, Egerton J, Bountra C, Williams NS, Anand P. Sensory fibres expressing capsaicin receptor TRPV1 in patients with rectal hypersensitivity and faecal urgency. Lancet. 2003 Feb 1;361(9355):385-91. doi: 10.1016/s0140-6736(03)12392-6. PMID 12573376
- [Background] Lewin GR, Mendell LM. Nerve growth factor and nociception. Trends Neurosci. 1993 Sep;16(9):353-9. doi: 10.1016/0166-2236(93)90092-z. PMID 7694405
- [Background] Anand P, Terenghi G, Warner G, Kopelman P, Williams-Chestnut RE, Sinicropi DV. The role of endogenous nerve growth factor in human diabetic neuropathy. Nat Med. 1996 Jun;2(6):703-7. doi: 10.1038/nm0696-703. PMID 8640566
- [Background] Micera A, Puxeddu I, Aloe L, Levi-Schaffer F. New insights on the involvement of Nerve Growth Factor in allergic inflammation and fibrosis. Cytokine Growth Factor Rev. 2003 Oct;14(5):369-74. doi: 10.1016/s1359-6101(03)00047-9. PMID 12948520
- [Background] Anand P, Pandya S, Ladiwala U, Singhal B, Sinicropi DV, Williams-Chestnut RE. Depletion of nerve growth factor in leprosy. Lancet. 1994 Jul 9;344(8915):129-30. doi: 10.1016/s0140-6736(94)91316-1. No abstract available. PMID 7912365
- [Background] Indo Y. Genetics of congenital insensitivity to pain with anhidrosis (CIPA) or hereditary sensory and autonomic neuropathy type IV. Clinical, biological and molecular aspects of mutations in TRKA(NTRK1) gene encoding the receptor tyrosine kinase for nerve growth factor. Clin Auton Res. 2002 May;12 Suppl 1:I20-32. doi: 10.1007/s102860200016. PMID 12102460
- [Background] March JS, Parker JD, Sullivan K, Stallings P, Conners CK. The Multidimensional Anxiety Scale for Children (MASC): factor structure, reliability, and validity. J Am Acad Child Adolesc Psychiatry. 1997 Apr;36(4):554-65. doi: 10.1097/00004583-199704000-00019. PMID 9100431